CLINICAL TRIAL: NCT05923125
Title: A Pilot Study of Pro-rEsolving and pRo-inflammatory reSPonses to Acute exhaustIve exeRcisE in Healthy Individuals
Brief Title: Pro-rEsolving and pRo-inflammatory reSPonses to Acute exhaustIve exeRcisE in Healthy Individuals
Acronym: PERSPIRE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: NYU Langone Health (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 23-00421
Record Dates: First submitted 2023-06-20; First posted 2023-06-28 (Actual); Last update posted 2025-02-27 (Actual); Status verified 2024-09

CONDITIONS: Exercise
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Healthy Adults (Experimental): Participants engage in a maximal exercise test. Before and after this test, blood samples are collected. At a separate, optional control visit, blood samples are collected as during the exercise visit, but participants do not participate in an exercise protocol.
  Interventions: Behavioral: Graded-Intensity Treadmill Exercise Protocol

INTERVENTIONS:
Behavioral: Graded-Intensity Treadmill Exercise Protocol — The exercise protocol will be administered by the principal investigator or other trained study staff under the supervision of the PI in the stress testing laboratory of NYU Langone Health - Tisch Hospital. The exercise protocol duration will vary by participant, but is likely to be between 8 and 25 minutes in duration.

SUMMARY:
This is a study of the effects of acute, exhaustive exercise on pro-resolving and pro-inflammatory responses in healthy, trained and untrained adults.

DETAILED DESCRIPTION:
The study requires one visit (a second, optional visit may occur). At the visit, participants will have blood drawn at several time points and also perform an exhaustive bout of treadmill exercise. Differences in specialized pro-resolving lipid mediators (SPMs) and other measures of inflammation and resolution over time will be characterized.

ELIGIBILITY:
Inclusion Criteria:

* Willingness and ability to provide informed consent and participate in PRESPIRE
* Able to read and speak English adequately to provide informed consent and understand verbal and written instructions. (the diet and sleep questionnaires are not validated in languages other than English)
* BMI < 27kg/m2
* Untrained: self-reporting no more than 1 day per week of regular exercise (inclusive of walking >5,000 steps daily and commuting via bicycle).
* Trained: self-reporting at least 4 hours of aerobic exercise / moderate or greater intensity physical activity weekly for the past year.

Exclusion Criteria:

* Anti-platelet medication use
* Chronic inflammatory or connective tissue disease
* History of bleeding or clotting disorder
* Immunological deficiency
* Diabetes mellitus
* Stage 2 or greater hypertension on screening
* Cardiovascular disease
* Chronic obstructive lung disease
* Anemia (hemoglobin <13g/dL in males or < 12 g/dL in females)
* Active smoking
* >5% body weight change over the past 6 months or plan to gain/lose weight during the study
* Platelet count <100,000
* Use of omega-3 fatty acid supplementation within 3 weeks of study participation
* Use of drugs or supplements known to inhibit COX-1/COX-2/lipoxygenases
* Corticosteroid use
* Use of beta-blocker medications
* Use of alpha-blocker medications
* Use of NSAIDs or aspirin within 2 weeks of study participation
* Vaccination within 2 weeks of study participation
* Pregnancy (a state of relative immunological deficiency)
* Any other cardiovascular, pulmonary, orthopedic, neurologic, psychiatric or other conditions that, in the opinion of the local clinician, would preclude participation and successful completion of the protocol.
* Any other illnesses that, in the opinion of the local clinician, would negatively impact or mitigate participation in and completion of the protocol

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 103 (Actual)
Dates: Start 2023-10-30 (Actual); Primary Completion 2025-01-29 (Actual); Study Completion 2025-01-29 (Actual)

PRIMARY OUTCOMES:
Change in Circulating Level of SPMs | Pre-Exercise, 4.5 Hours Post-Exercise (Day 1)
  Circulating level (%) of serum, plasma and neutrophil (SPMs) will be measured using patient blood draws.
  Circulating level of SPMs is calculated as a composite endpoint.

CONTACTS AND LOCATIONS:
Overall Officials: Sean P. Heffron, MD, Principal Investigator — NYU Langone Health
Locations (1):
- Tisch Hospital, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No
Data sharing will be considered, however the study team does not anticipate data will be made public outside of publication.